CLINICAL TRIAL: NCT06112236
Title: Effects of Treatments for Anemia and Iron Deficiency on the Electrolyte Balance in Lung Transplant Recipients: A Special Focus on Hypophosphatemia
Status: Active, not recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-02302
Record Dates: First submitted 2023-06-27; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Hypophosphatemia
MeSH Terms: conditions — Hypophosphatemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The aim of this study is to generate evidence regarding hypophosphatemia after iron infusion in lung transplant recipients in context of anemia and/or iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

* lung transplant recipient
* treated at the University Hospital Zurich between 2015 until 2022

Exclusion Criteria:

* Denied general consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lung transplant recipient
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of serum phosphate level | Baseline and up to 90 days after iron infusion
  Change of serum phosphate level before and after iron infusion

SECONDARY OUTCOMES:
Change of urin phosphate level | Baseline and up to 90 days after iron infusion
  Change of urin phosphate level before and after iron infusion
Change of hemoglobin | Baseline and up to 90 days after iron infusion
  Change of hemoglobin level before and after iron infusion
Change of mean corpuscular volume (MCV) | Baseline and up to 90 days after iron infusion
  Changes of serum MCV level before and after iron infusion
Change of mean corpuscular hemoglobin (MCH) | Baseline and up to 90 days after iron infusion
  Change of serum MCH level before and after iron infusion
Change of serum magnesium | Baseline and up to 90 days after iron infusion
  Change of serum magnesium level before and after iron infusion
Change of serum and urin calcium | Baseline and up to 90 days after iron infusion
  Change of serum and urin calcium level before and after iron infusion
Change of serum albumin | Baseline and up to 90 days after iron infusion
  Change of serum albumin level before and after iron infusion
Complications after iron infusion | 2015-2022
  Number of patients with complications due to hypophosphatemia after iron infusion (Hospitalization, hypoxia, fracture due to hypophosphatemia)
Predictors | baseline and up to 90 days after iron infusion
  Analysis of possible predictors for the decrease of serum phosphate levels after iron infusion
Therapeutic management | 2015 to 2022
  Descriptive analysis of therapeutic management of hypophosphatemia after iron infusion

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided